CLINICAL TRIAL: NCT05378776
Title: Triage Administration of Sucrose for Gastroenteritis in Children; a Randomized Controlled Trial
Brief Title: Sucrose at Triage for Acute Gastroenteritis Episode in Children
Acronym: STAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jocelyn Gravel (Other)
Responsible Party: Sponsor-Investigator, Jocelyn Gravel, Principal investigator, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-4319
Record Dates: First submitted 2022-05-06; First posted 2022-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Gastroenteritis Acute; Vomiting
Keywords: children; sucrose; emergency department; triage
MeSH Terms: conditions — Vomiting; Emergencies | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: It is a blinded study for participants, treating physician and statistician. However, for practical reasons and to minimize cost related to the study preparation, the research nurses/assistants will not be blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucrose (Experimental): The experimental arm will receive 1.5 ml/kg of the sucrose solution at triage (once). The composition of the homemade sucrose solution used in our emergency department is 3.5 g of table sugar (sucrose) mixed with 10 ml of diluted juice (see standard arm description) to obtain a solution with the same appearance as the standard arm.
  Interventions: Dietary Supplement: sucrose
- Control (Placebo Comparator): This group will receive 1.5 mL/kg of diluted juice composed of juice (apple or orange) and water in equal proportion once at triage. This solution contains 0.05 g/ml of sucrose for a total of 0.075 g/kg of sucrose (eight times less than the intervention arm).
  Interventions: Dietary Supplement: Standard rehydration solution

INTERVENTIONS:
Dietary Supplement: sucrose — The experimental arm will receive 1.5 ml/kg of the sucrose solution at triage (once). The composition of the homemade sucrose solution used in our emergency department is 3.5 g of table sugar (sucrose) mixed with 10 ml of water. For this double-blind study, we replaced water with diluted juice (see standard arm description) to obtain a solution with the same appearance as the standard arm. With the idea of correcting ketosis, we chose to provide the same amount of sugar as we do in hypoglycemia (0.4-0.5 g/kg of dextrose) to participants in the intervention group, which represents 1.5 ml/kg of the sucrose solution containing 0.4 g of sucrose/mL for a total of 0.6 g/kg of sucrose.
  Arms: Sucrose
Dietary Supplement: Standard rehydration solution — This group will receive 1.5 mL/kg of diluted juice composed of juice (apple or orange) and water in equal proportion once at triage. This solution contains 0.05 g/ml of sucrose for a total of 0.075 g/kg of sucrose (eight times less than the intervention arm).
  Arms: Control

SUMMARY:
Background: Acute viral gastroenteritis is a very common pediatric medical condition that results in a large number of emergency department (ED) visits. Fasting-induced ketosis has been suggested to contribute to nausea and vomiting in children with VGE. To date, there is no data on the impact of oral sucrose intake during oral rehydration.

Objective: The aim of this study is to assess the impact of providing a sucrose solution at triage to young children with suspected acute viral gastroenteritis on the amount of rehydration solution intake in the first 2 hours. We will also assess the proportion of discharge after initial medical evaluation, the proportion of oral rehydration failure, the number of vomiting episodes per patient, ondansetron administration, the time between the intervention and ED discharge, the time between the first medical contact and ED discharge and return visits within 48 hours.

Methods:

This study will be a double-blind randomized controlled trial. Recruitment will take place in a tertiary pediatric ED. Participants will be all children who present to the ED with suspected acute acute viral gastroenteritis with at least three vomiting in the previous 24 hours. The intervention will consist in giving 1.5 ml/kg of a sucrose solution composed of diluted juice with added table sugar (3.5g of sucrose/10 ml) compared with 1.5 ml/kg of diluted juice (0.5g of sucrose/10 mL, standard of care in our ED). Following that, all participants will be rehydrated with 15 mL of diluted juice every 15 minutes or more if tolerated. The primary outcome will be the amount of rehydration solution (ml) absorbed in the first two hours following intervention. Secondary outcomes will include disposition after initial medical evaluation, oral rehydration failure, the number of vomiting, ondansetron administration, the time between the intervention and ED discharge, the time between the first medical contact and ED discharge and return visits within 48 hours. The primary analysis will be the difference in the amount of tolerated oral rehydration between the two groups. Based on a preliminary study of children suffering from VGE, it was estimated that the recruitment of 238 participants would provide a power of 80% to identify a difference of 15 ml between the two groups.

Expected results:

We hope that this study will demonstrate that an oral sucrose solution given at triage to children presenting with symptoms compatible with acute acute viral gastroenteritis promotes oral hydration and consequently increases the total amount of rehydration solution tolerated by children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 6 years. We will restrict to this age group to have a more homogenous group.
* At least 3 non-bilious, non-bloody, vomiting in the last 24 hours
* No other diagnostic more likely than acute viral gastroenteritis suspected at triage

Exclusion Criteria:

* Severe dehydration (based on poor capillary refill or hypotension)
* Hypoglycemia identified by the triage nurse (< 2,8 mmol)
* Bilious or bloody vomiting
* Chronic disease other than asthma
* Previous inclusion in the study
* Inability to obtain parental informed consent (language barrier, absence, etc.)

Ages: 6 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mean amount of tolerated oral rehydration in mL | 2 hours after intervention
  The total amount of rehydration solution tolerated during the two hours following intervention. This will be the amount of solution absorbed by the child without vomiting. In case of vomiting, the amount of solution absorbed will be the amount of solution tolerated after vomiting. In the few situations when the children will be discharged from the ED before two hours, we will collect the amount of solution tolerated before discharge.

SECONDARY OUTCOMES:
Number of participants who needed an observation | 2 hours
  Patient who are not immediately discharged by the treating physician after the first evaluation
Number of participants with oral rehydration failure | 6 hours
  Patient who need an intravenous rehydration during ED stay
Mean number of vomiting | 6 hours
  Number of vomiting episode per patient during ED stay
Number of participants who received ondansetron | 6 hours
  Number of patients who received ondansetron during ED stay
Mean length of stay | 24 hours
  The time between the intervention and ED discharge
Mean length of stay after physician evaluation | 24 hours
  The time between the first evaluation by a physician and ED discharge
Number of participants who had a return visit | 48 hours
  return visit to the ED

CONTACTS AND LOCATIONS:
Locations (1):
- Sainte-Justine Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided